CLINICAL TRIAL: NCT03823833
Title: Systematic Proposal of Fertility Preservation by Oocyte Freezing in Case of Benign Ovarian Tumors With High Risk of Recurrence
Brief Title: Oocyte Freezing for Fertility Preservation in Benign Ovarian Tumors
Acronym: OFBOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_48
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis; Dermoid Cyst; Mucinous Cyst
Keywords: Oocyte freezing; fertility preservation; ovarian cysts; benign ovarian tumor; endometrioma
MeSH Terms: conditions — Endometriosis; Dermoid Cyst; Mucocele; Ovarian Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Benign ovarian cysts are frequent during women's life. They are diagnosed with pelvic pain or fortuitously during an ultra-sonographic exam. In case of persistence,a surgery will be necessary to identify the nature of the cyst and assess its benignity. In some case, cysts are recurrent and multiple surgeries are needed leading to a significant risk of ovarian damage by follicular depletion. Oocyte cryopreservation is no longer considered as an experimental technique of Fertility Preservation since 2013 as it has been recognized to be efficient and safe. According to reproductive medicine scientific committees and the French ethic law, fertility preservation has to be proposed in every situation of infertility risk. To date, there is no cohort study dedicated to fertility preservation by oocyte freezing in this specific subgroup of patients. The purpose of the study is to prospectively evaluate the oocyte number and quality after controlled ovarian hyperstimulation in patients with recurrent ovarian cysts.

ELIGIBILITY:
Inclusion Criteria:

* women with benign ovarian tumor with high risk of recurrence, i-e, endometrioma, dermoid cysts or mucinous cysts.
* women with previous surgery and/or high risk of ovarian damage: bilateral cysts, cyst diameter higher than 5 cms
* Having a social insurance
* Able to give an informed consent

Exclusion Criteria:

* Borderline tumors
* Undetectable AMH levels
* Personal history of thrombo-embolic events
* pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — young women
Study Population: Young women with benign ovarian tumors and high risk of further infertility due to surgery
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes eligible for cryopreservation | After 15 days of controlled ovarian hyperstimulation (COH)

SECONDARY OUTCOMES:
Percentage of immature or morphologically abnormal oocytes | Real-time, the day of egg retrieval
Number of mature follicles (≥15 mm) and intermediary (10-14 mm) during ovarian stimulation | The day of HCG triggering at the end of ovarian stimulation
Questionnaire on tolerance and complications | One week after the egg retrieval
  A systematic telephone interview will be carried out 48 to 72 hours after the oocyte puncture to judge the tolerance of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Decanter, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France